CLINICAL TRIAL: NCT01696669
Title: Phase 2, Open-label, Uncontrolled, Multicenter and Prospective Study of Intensive Chemotherapy, Surgery and Radiotherapy to Treat Ewing's Sarcoma in Children and Young Adults
Brief Title: Study of Intensive Chemotherapy, Surgery and Radiotherapy to Treat Ewing's Sarcoma in Children and Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Principal Investigator, Mariló de Carrillo, Jaume Mora, Grupo Espanol de Investigacion en Sarcomas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS-21; 2009-016027-62 (EudraCT Number)
Record Dates: First submitted 2011-06-30; First posted 2012-10-01 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Ewing's Sarcoma
Keywords: Ewing's Sarcoma; P6 protocol MSKCC; Gemcitabine; Docetaxel
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Drug Therapy; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy + Surgery + Radiotherapy (Experimental): Standard risk patients: MP6 Treatment:
  CHEMOTHERAPY: 2 cycles of vincristine-doxorubicin + dexrazoxane-cyclophosphamide, 1 cycle of ifosfamide-etoposide. SURGERY: Ideally within 21 days after chemotherapy.
  CHEMOTHERAPY: 1 cycle of vincristine-doxorubicin + dexrazoxane-cyclophosphamide, 1 cycle of ifosfamide-etoposide.
  RADIOTHERAPY: On the primary tumor bed in case of unresectable tumors, resected tumors with inadequate margins, or those with histologic response <90%.
  High risk patients:
  CHEMOTHERAPY: Window phase with 2 cycles of gemcitabine + docetaxel. MP6 TREATMENT. CHEMOTHERAPY: Maintenance therapy for 1 year with gemcitabine + docetaxel.
  Interventions: Drug: Chemotherapy; Procedure: Surgery; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Chemotherapy — * Vincristine, 2 mg/m^2 IV bolus, day 1.
  * Doxorubicin: 75 mg/m^2 per cycle, or 25 mg/m^2/day x 3 days, IV infusion, 1 hour (after dexrazoxane administration at the dose of 10:1).
  * Dexrazoxane: administered at a dose of 10:1, before doxorubicin only in adults.
  * Cyclophosphamide: 2100 mg/m^2 IV infusion, 6 hours, with MESNA protection, days 1 and 2.
  * MESNA: used with cyclophosphamide and ifosfamide. The total daily dose of MESNA is equivalent to at least 60% of the daily dose of cyclophosphamide or ifosfamide.
  * G-CSF: 5 micrograms/kg/day SC. It starts 24 hours after the last dose of chemotherapy and continues until the absolute neutrophil count is ≥ 750 mm^3/L.
  * Ifosfamide: 1800 mg/m^2/day IV infusion, 1 hour, days 1-5 of each cycle (9,000 mg/m^2 total maximum dose).
  Window phase in high-risk patients (21-days cycle):
  * Gemcitabine: 1000 mg/m^2 IV, 90 minutes on day 1 and 8.
  * Docetaxel 100 mg/m^2, 2-3 hour infusion on day 8.
Procedure: Surgery — Surgical intervention aiming to completely resect the tumor with negative margins.
Radiation: Radiotherapy — On the primary tumor bed in case of unresectable tumors, resected tumors with inadequate margins, or those with histologic response <90%. Patients will receive radiotherapy 21 days after the completion of chemotherapy.

SUMMARY:
Tumors of the Ewing sarcoma family (ES) affect children, adolescents and young adults. The reported incidence is 0.6 cases per million inhabitants every year. The peak incidence occurs between 10 and 20 years and it is rarely diagnosed beyond 30. The ES is a severe disease with a progression-free survival after 5 years of 60% in cases without metastasis and deadly in the majority of patients presenting metastasis. The ES is considered a systemic disease because, despite receiving an adequate local treatment, over 90% of patients deaths occur due to disseminated disease. Combined therapy of surgery, radiotherapy and chemotherapy has led to an improvement in the prognosis, achieving a survival of about 60% in most series

The MSKCC P6 protocol was developed for the treatment of high risk ES. In 2003, Kolb et al. reported the MSKCC experience after a 4-years follow-up of 68 patients who had been included from 1990 to 2001. Following the MSKCC P6 protocol, a survival rate of 82% was achieved in patients without metastasis, superior to the achieved with less intensive protocols. Following the guidelines of the MSKCC P6 protocol, in 2002 we modified the treatment schedule to create the modified P6 protocol (MP6). GEIS intends to develop MP6 as a clinical trial, which could provide the following potential advantages about current treatments:

1. Lower total dose of alkylating agents.
2. Early cardioprotection with dexrazoxane.
3. Radiotherapy adjusted to the initial response.
4. Pilot trial with the combination of Gemcitabine + Docetaxel for high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ewing's Sarcoma in which the molecular analysis has been performed in one of the 2 reference laboratories of the study and the EWS gene rearrangement has been confirmed by RT-PCR in the Hospital Sant Joan de Déu de Barcelona, or by fluorescence in situ hybridization (FISH) in the Cancer Research Center of Salamanca.
* High-risk patients will be those patients with metastases, patients with primary tumor in pelvis or axial bones and patients with (micro) metastases in bone marrow detected by the molecular study. The remaining patients will be considered as standard risk. Lung nodules identified by CT-scan with diameter > 5 mm will be considered metastatic. Nodules ≤ 5 mm will be biopsied.
* Age ≤ 40 years.
* Adequate renal and hepatic function , defined as calculated creatinine clearance > 60 ml/min, creatinine, total bilirubin, AST and/or ALT < 1,5 times the upper limit of normal (ULN).
* Normal cardiac function defined by echocardiography, or ejection fraction ≥ 55%.
* ECOG performance status 0 - 1 (Appendix VIII).
* Informed consent form signed by parents, guardians or the patient (if over 18 years), prior to the start of treatment.
* Patients of childbearing age (both men and women) must use effective contraceptive methods before study entry and during the realization of it. Effective contraceptive methods for both women and men should be extended to 6 months after stopping the treatment under study. Pregnancy must be excluded by urine test (negative pregnancy test) prior to the inclusion in the study.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Active infection or other severe concomitant diseases.
* Severe psychiatric conditions that make impossible to obtain the signed informed consent form or limit the treatment compliance.
* Concurrent treatment with other experimental drugs within 30 days prior to study entry.
* History of previous cancer diagnosed or treated in the past 5 years except basal cell carcinoma, cervical carcinoma in situ or superficial bladder cancer.

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2010-03-30 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Assessment of the progression free survival in all the patients enrolled in the study 3 years after the completion of the treatment under study.
  Assessment of the progression free survival in all the patients enrolled in the study 3 years after the completion of the treatment under study.

SECONDARY OUTCOMES:
Objective response rate (ORR) | two months
  To assess the objective response rate to treatment (ORR) defined following EMEA criteria (CPMP/EWP/205/95/Rev.3/Corr.2) in high risk patients with Ewing's sarcoma treated with an early window phase of Gemcitabine + docetaxel (G + D).
Assessment of disease progression | to reach an index of disease progression < 20% for high risk patients during the maintenance phase with Gemcitabine + Docetaxel.
  To assess the disease progression, aiming to reach an index of disease progression < 20% for high risk patients during the maintenance phase with Gemcitabine + Docetaxel.
evaluate the toxicity and tolerance to the treatment Gemcitabine + Docetaxel in high risk patients, and toxicity and tolerance of mP6 treatment in all patients. | 12 months
  To evaluate the toxicity and tolerance to the treatment Gemcitabine + Docetaxel in high risk patients, and toxicity and tolerance of mP6 treatment in all patients.
Assessment of bone marrow condition. | 24 months
  Molecular diagnosis and extension study of bone marrow in all patients included in the trial. Assessment of prognostic significance of the type of translocation and the molecular effect in the bone marrow.
Study the impact of patients treated with Cardioxane in cardioprotection | 6 months
  Creation of a cohort of patients treated with anthracyclines at high doses and early cardioprotection with dexrazoxane (Cardioxane). Long-term study of cardioprotection in these patients compared with historical series from the P6 protocol that did not received cardioprotection.

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Mora Graupera, MD, Study Chair — GEIS
Locations (9):
- Spain (9):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Institut Català d'Oncologia l'Hospitalet, L'Hospitalet de Llobregat
  - Hospital Ramón y Cajal, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Miguel Servet, Zaragoza